CLINICAL TRIAL: NCT01004887
Title: Diagnostic And Prognostic Markers In High-Grade Glioma
Brief Title: Study of Tissue and Blood Samples From Patients With High-Grade Glioma
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCCTG-94-72-52; NCCTG-947252; CDR0000406625 (Registry Identifier: PDQ (Physician Data Query)); NCI-2009-00688 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma; childhood high-grade cerebellar astrocytoma; childhood high-grade cerebral astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Glioblastoma; Gliosarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood and tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group: Patients with newly diagnosed high-grade gliomas participating in NCCTG/Alliance or Mayo protocols. Previously collected blood and tissue samples are analyzed via PCR, IHC, flow cytometry, and FISH.
  Interventions: Other: diagnostic laboratory biomarker analysis

INTERVENTIONS:
Other: diagnostic laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at tissue and blood samples from patients with high-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the diagnostic and prognostic relevance of various molecular, cytogenetic, and other tumor markers in high-grade glioma in paraffin-embedded tissue collected from patients enrolled in the Mayo Clinic or North Central Cancer Treatment Group (NCCTG) high-grade glioma trials conducted since 1979.
* To evaluate alterations of specific chromosomes and chromosomal regions including 7, 9p, 10p, 10q, 13q, 17p, 17q, 19q, 22q, X, and Y using PCR analysis of microsatellite repeats and FISH.
* To determine DNA ploidy by flow cytometric analysis.
* To examine various markers of cellular proliferation and cellular function including flow cytometric determination of %S-phase, %G2M, and immunohistochemical evaluation of PCNA, Ki-67, and p53.
* To evaluate additional markers identified by the Glioma Markers Network.
* To compare the incidence of markers in the major histologic subtypes (anaplastic astrocytoma [AA], anaplastic oligoastrocytoma [AOA], glioblastoma multiforme [GBM]) and to assess their correlation in the total group, as well as within each of these subtypes.
* To compare the ploidy determinations by FISH and flow cytometry.

OUTLINE: Paraffin-embedded tissue and peripheral blood samples, previously or currently collected from clinical trials participants at the time she/he enrolled in the trial, are evaluated for as many markers as possible, changes in cytogenic and molecular genetic tumor markers, frequency distributions of all tumor markers and histological and clinical variables by polymerase chain reaction, IHC, flow cytometry, and FISH analysis.

ELIGIBILITY:
* Patients with newly diagnosed high-grade gliomas
* Patients participating in NCCTG/Alliance or Mayo protocols
* Willing to provide mandatory blood and tissue samples for research purposes; note: 15 unstained slides may be submitted in place of a tissue block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed high-grade gliomas participating in NCCTG/Alliance or Mayo protocols.
Sampling Method: Probability Sample
Enrollment: 631 (Actual)
Dates: Start 1995-11 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
time to progression | baseline
survival | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jan Buckner, MD, Study Chair — Mayo Clinic
Locations (110):
- United States (110):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia